CLINICAL TRIAL: NCT05031117
Title: Comparative Study Between Dural Puncture Epidural Technique and Conventional Epidural Technique During Laparoscopic Assisted Vaginal Hysterectomy
Brief Title: Dural Puncture Epidural Technique For Vaginal Procedures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Reham Ali Abdelhaleem Abdelrahman, Anesthesia lecturer M.D., Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: ZO-19251
Record Dates: First submitted 2021-08-28; First posted 2021-09-01 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Gynecologic Diseases Requiring Vaginal Hysterectomy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Epidural Technique (Experimental)
  Interventions: Procedure: 25G Dural Puncture Epidural Technique
- Dural Puncture Epidural technique using pencil-point 25G Whitacre needle (Active Comparator)
  Interventions: Procedure: Conventional Epidural Technique

INTERVENTIONS:
Procedure: Conventional Epidural Technique — Standard Lumbar Epidural Technique at L4-5 interspace using Tuhoy needle (18G) then epidural catheter (20G) inserted, then 15ml 0.5% Bupivacane and 50ug fentanyl given.
  Arms: Dural Puncture Epidural technique using pencil-point 25G Whitacre needle
Procedure: 25G Dural Puncture Epidural Technique — 25G pencil point spinal needle will be inserted at L4-5 interspace through the tuhoy needle
  Arms: Conventional Epidural Technique

SUMMARY:
25G Dural Puncture Epidural Technique will be compared with Conventional Standard Lumbar Epidural Technique During Anesthesia of Laparoscopic Assisted Vaginal Hysterectomy.

ELIGIBILITY:
Inclusion Criteria:

* Age: 25-55 years old.
* Height: 165 cm.

Exclusion Criteria:

* Patient Refusal.
* Coagulopathy.
* Deformity of lumbar vertebrae.

Ages: 25 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2022-01-10 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2023-02-19 (Actual)

PRIMARY OUTCOMES:
incidence of bilateral sacral blockade | Up to 30 minutes after local anesthetic injection

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesia, Surgical ICU, and Pain Management, Cairo, Egypt